CLINICAL TRIAL: NCT02357576
Title: Phase 3 Study of Standard Lipid Therapy Versus Intravenous Fat Emulsion Minimization for the Prevention of Parenteral Nutrition-Associated Liver Disease
Brief Title: Standard Lipid Therapy vs IVFE Minimization for Prevention of PNALD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Seattle Children's Hospital (Other); University of Florida (Other); Primary Children's Hospital (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Meghan A. Arnold, MD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00075458; 1R01FD005085-01A1 (FDA)
Record Dates: First submitted 2015-02-02; First posted 2015-02-06 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cholestasis
MeSH Terms: conditions — Cholestasis | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced Lipid (Experimental): Subjects will receive a minimized dose (1 g/kg/day) of the soybean-based lipid component of parenteral nutrition.
  Interventions: Drug: Intralipid 20% I.V. Fat Emulsion
- Standard Lipid (Active Comparator): Subjects will receive the standard dose (up to 3 g/kg/day) of the soybean-based lipid component of parenteral nutrition.
  Interventions: Drug: Intralipid 20% I.V. Fat Emulsion

INTERVENTIONS:
Drug: Intralipid 20% I.V. Fat Emulsion

SUMMARY:
Parenteral nutrition-associated cholestasis (PNAC) and liver disease (PNALD) are associated with significant morbidity and mortality in neonates and is felt to be exacerbated by soybean-based lipid emulsions. Much research is currently being directed at identifying ways to reduce this risk. Reduction of the dose of soybean-based lipid given as a component of parenteral nutrition is one possible strategy. In this study we will compare standard dosing of soybean-based lipid (up to 3/kg/day) with a minimized dose (1 g/kg/day) and evaluate for the development of cholestasis and adequate growth between the two groups. Longterm followup will include an assessment of neurodevelopmental outcomes at 12 and 24 months of age.

Funding source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* neonates and infants who are at least 28 weeks corrected gestational age at the time of enrollment who are parenteral nutrition (PN) naive
* current direct bilirubin <2 mg/dL
* any of the following conditions:
* meconium ileus and peritonitis
* gastroschisis
* omphalocele >4cm or with liver herniated outside of the abdominal cavity
* necrotizing enterocolitis requiring surgical intervention
* volvulus
* intestinal atresia with >50% bowel loss

Exclusion Criteria:

* weight <1 kg
* metabolic pathway defect which is associated with liver dysfunction in the neonatal period, including: hereditary fructose intolerance, galactosemia due to transferase deficiency and neonatal tyrosinemia, and/or disorder of lipid metabolism
* hepatic insufficiency as documented by either a biopsy with cirrhosis and/or marked aberration in synthetic function
* renal failure
* primary or secondary liver disease, regardless of liver function (includes hepatitis)
* use of extracorporeal membrane oxygenation (ECMO)
* suspected congenital obstruction of the hepatobiliary tree
* documented active infection which may be communicable, including infections hepatitis or HIV
* previous receipt of choleretic agents
* currently receiving phenobarbital or other barbiturates
* history of PNAC
* direct bilirubin >=2 mg/dL at time of enrollment
* congenital or acquired anomaly which will require major cardiovascular surgery
* major congenital or chromosomal anomaly
* hypoxic ischemic encephalopathy
* congenital defect of the brain
* major seizure disorder

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2016-05-21 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan A Arnold, MD, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - University of Colorado/Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who were enrolled were randomized shortly after enrollment. 1 patient was removed immediately after enrollment, before intervention, due to a screen fail.
Groups:
- Reduced Lipid: Subjects will receive a minimized dose (1 g/kg/day) of the soybean-based lipid component of parenteral nutrition.
  Intralipid 20% I.V. Fat Emulsion
- Standard Lipid: Subjects will receive the standard dose (up to 3 g/kg/day) of the soybean-based lipid component of parenteral nutrition.
  Intralipid 20% I.V. Fat Emulsion
Period: Treatment Period
Arm/Group | Reduced Lipid | Standard Lipid
Started | 12 | 9
Completed | 12 | 7
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Neurodevelopmental Outcome Follow Up
Arm/Group | Reduced Lipid | Standard Lipid
Started | 11 (1 patient exited the study after treatment completion and before returning for follow up visits.) | 7
Completed (Completed 24 Month Follow Up) | 6 | 2
Not Completed | 5 | 5
Not completed — Scheduling error | 1 | 1
Not completed — Became ineligible during follow-up | 1 | 0
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Lipid | Standard Lipid | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: days] — Age at randomization in TATUM
  days | 2 [0 to 4] | 2 [1 to 4] | 2 [0 to 4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 8 | 5 | 13
  Other | 0 | 1 | 1
  Unknown | 0 | 2 | 2
Diagnosis [Count of Participants; unit: Participants]
  Gastroschisis | 12 | 8 | 20
  Intestinal atresia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Rise of Direct Bilirubin as a Function of Time
Description: The rate of rise (change over time) of direct bilirubin was compared between the two groups at different time points.
Time Frame: 12 weeks
Population: Analyzable data was not available for one participant in the Reduced Lipid Arm
Measure: Number (95% Confidence Interval); unit: mg/dL/day
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 11 | 9
mg/dL/day
  1 Day from Baseline | 1.033001353 [1.011427197 to 1.055035694] | 1.05457485 [1.029533513 to 1.080225375]
  7 Days from Baseline | 1.025504411 [1.005132124 to 1.046289609] | 1.049318179 [1.025241711 to 1.07396016]
  28 Days from Baseline | 0.999691048 [0.981391909 to 1.018331496] | 1.031125269 [1.008439715 to 1.05432115]
  56 Days from Baseline | 0.96628119 [0.945472667 to 0.987547779] | 1.007357736 [0.981844238 to 1.033534209]
  84 Days from Baseline | 0.933987896 [0.907126199 to 0.961645019] | 0.984138047 [0.952398442 to 1.016935507]

2. Secondary Outcome: Prevalence of Parenteral Nutrition-associated Cholestasis (PNAC) (Direct Bilirubin ≥2 mg/dL)
Description: The number of participants who had a direct bilirubin ≥2 mg/dL were compared between the standard and reduced lipid groups. Bilirubin data was collected from baseline until 7 days after PN has been discontinued, but not to exceed a total of 12 weeks.
Time Frame: 12 weeks
Population: Analyzable data was not available for one participant in the Reduced Lipid Arm
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 11 | 9
Participants | 2 | 3
Statistical Analysis 1: Comparison: Reduced Lipid vs Standard Lipid; Test type: Other — Percentage and frequencies were used to describe the incidence of PNAC in the two groups; p = 0.617, Fisher Exact

3. Secondary Outcome: Prevalence of Severe Parenteral Nutrition-associated Cholestasis (PNAC) (Direct Bilirubin ≥4 mg/dL in Subjects on Parenteral Nutrition for at Least 2 Weeks)
Description: The number of participants with severe PNAC defined as a direct bilirubin ≥4 mg/dL were compared between the standard and reduced lipid groups. Bilirubin data was collected from baseline until 7 days after PN has been discontinued, but not to exceed a total of 12 weeks.
Time Frame: 12 weeks
Population: Analyzable data was not available for one participant in the Reduced Lipid Arm
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 11 | 9
Participants | 0 | 1
Statistical Analysis 1: Comparison: Reduced Lipid vs Standard Lipid; Test type: Other — Percentage and frequencies were used to describe the incidence of severe PNAC; p = 0.450, Fisher Exact

4. Secondary Outcome: The Time to Development of PNAC
Description: The time to development was compared between the standard and reduced lipid groups.
Time Frame: 12 weeks
Population: Only the subjects that developed PNAC were analyzed
Measure: Median (Full Range); unit: days
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 2 | 3
days | 19.50 [14 to 25] | 39.00 [29 to 42]
Statistical Analysis 1: Comparison: Reduced Lipid vs Standard Lipid; Test type: Other — The Kaplan Meier curve was used to evaluated the time to first PNAC event; p = 0.2716, Log Rank; A log rank test was used to test the equality of the survival curve between the two groups

5. Secondary Outcome: The Time to Development of Severe PNAC
Description: The time to development from randomization was compared between the standard and reduced lipid groups.
Time Frame: 12 weeks
Population: Subjects who developed severe PNAC as defined by a direct bilirubin value of 4 mg/dL or greater
Measure: Number; unit: Days
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 0 | 1
Days |  | 42

6. Secondary Outcome: Peak Total Bilirubin Level
Description: The peak (highest) total bilirubin collected from each subject from after week 1 to end of treatment. This was compared between the standard and reduced lipid groups.
Time Frame: 12 weeks
Population: Subjects with total bilirubin values collected after 1 week
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 12 | 9
mg/dL | 1.7 [0.2 to 9.9] | 2.9 [0.7 to 9.9]

7. Secondary Outcome: Peak Direct Bilirubin Level
Description: The peak (highest) direct bilirubin collected from each subject from after week 1 to end of treatment. This was compared between the standard and reduced lipid groups.
Time Frame: 12 weeks
Population: Subjects with direct bilirubin values collected after 1 week
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 11 | 8
mg/dL | 0.8 [0.3 to 2.5] | 1.7 [0.6 to 4]

8. Secondary Outcome: The Prevalence of Essential Fatty Acid Deficiency (EFAD)
Description: The number of participants who experienced EFAD was compared between the standard and reduced lipid groups.
Time Frame: 12 weeks
Population: All patients in the reduced lipid group were analyzed. The standard lipid group had essential fatty acid profile drawn for one patient as not all patients in the standard group required the essential fatty acid profile to be drawn.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 12 | 1
Participants | 2 | 0

9. Secondary Outcome: Adequacy of Growth as Evaluated by Z-scores for Weight
Description: Z-scores were compared between subjects in the two treatment groups by week. Z-scores are the number of standard deviations above (positive value) or below (negative value) the median on the FENTON and WHO growth charts. Fenton scores were used for infants born <37 weeks gestation. WHO scores were used for infants born at ≥37 weeks gestation.
Time Frame: 12 weeks
Population: All subjects aside from the screen fail. Z-scores were recorded while subjects were "on treatment" which meant that they were recorded until 7 days after parenteral nutrition (PN) had been discontinued, but not to exceed 12 weeks for subjects still on PN. This is why the participants analyzed each week is a different number and decreasing with time
Measure: Median (Full Range); unit: z-score
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 12 | 9
z-score
  Birth | -1.36 [-3.14 to 0.47] | -0.93 [-1.71 to 1.06]
  Study Week 1 | -2.28 [-3.46 to -0.3] | -1.85 [-2.26 to 0.65]
  Study Week 2: number analyzed (Participants) | 12 | 8
  Study Week 2 | -2.32 [-3.49 to -0.6] | -1.3 [-2.38 to -0.03]
  Study Week 3: number analyzed (Participants) | 11 | 6
  Study Week 3 | -2.33 [-3.73 to -0.59] | -1.485 [-2.47 to 0.44]
  Study Week 4: number analyzed (Participants) | 10 | 5
  Study Week 4 | -2.575 [-3.61 to -0.84] | -1.59 [-2.01 to -1.19]
  Study Week 5: number analyzed (Participants) | 9 | 3
  Study Week 5 | -2.42 [-3.52 to -0.44] | -1.78 [-2.34 to -1.04]
  Study Week 6: number analyzed (Participants) | 7 | 3
  Study Week 6 | -2.54 [-3.81 to -0.55] | -1.88 [-2.49 to -0.89]
  Study Week 7: number analyzed (Participants) | 5 | 2
  Study Week 7 | -2.37 [-3.48 to -0.28] | -1.62 [-2.53 to -0.71]
  Study Week 8: number analyzed (Participants) | 4 | 2
  Study Week 8 | -1.86 [-2.66 to -0.55] | -1.745 [-2.68 to -0.81]
  Study Week 9: number analyzed (Participants) | 3 | 2
  Study Week 9 | -2.25 [-2.38 to -0.41] | -1.745 [-2.46 to -1.03]
  Study Week 10: number analyzed (Participants) | 2 | 2
  Study Week 10 | -1.415 [-2.44 to -0.39] | -1.785 [-2.55 to -1.02]
  Study Week 11: number analyzed (Participants) | 2 | 2
  Study Week 11 | -1.355 [-2.31 to -0.4] | -1.885 [-2.41 to -1.36]
  Study Week 12: number analyzed (Participants) | 2 | 2
  Study Week 12 | -1.33 [-2.36 to -0.3] | -1.885 [-2.56 to -1.21]

10. Secondary Outcome: Adequacy of Growth as Evaluated by Z-scores for Height
Description: Z-scores were compared between subjects in the two treatment groups. Z-scores are the number of standard deviations above (positive value) or below (negative value) the median on the FENTON and WHO growth charts. Fenton scores were used for infants born <37 weeks gestation. WHO scores were used for infants born at ≥37 weeks gestation.
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Median (Full Range); unit: z-score
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 12 | 9
z-score
  Birth | -1.06 [-3.84 to 0.29] | -0.87 [-2.62 to 1.12]
  Study Week 1 | -1.365 [-4.41 to 0] | -1.22 [-3.2 to 0.96]
  Study Week 2: number analyzed (Participants) | 11 | 8
  Study Week 2 | -1.53 [-4.22 to -0.58] | -1.55 [-3.73 to 0.21]
  Study Week 3: number analyzed (Participants) | 11 | 6
  Study Week 3 | -2.19 [-4.77 to -0.65] | -1.775 [-2.57 to 0.56]
  Study Week 4: number analyzed (Participants) | 10 | 5
  Study Week 4 | -2.15 [-4.6 to -0.56] | -1.91 [-2.72 to 0.06]
  Study Week 5: number analyzed (Participants) | 8 | 3
  Study Week 5 | -3.21 [-4.57 to -0.28] | -2.11 [-3.25 to -1.48]
  Study Week 6: number analyzed (Participants) | 7 | 3
  Study Week 6 | -1.81 [-4.52 to -0.13] | -2.37 [-3.25 to -1.14]
  Study Week 7: number analyzed (Participants) | 5 | 2
  Study Week 7 | -1.56 [-3.37 to -0.98] | -2.39 [-3.47 to -1.31]
  Study Week 8: number analyzed (Participants) | 4 | 2
  Study Week 8 | -0.98 [-1.71 to 2.93] | -2.51 [-3.29 to -1.73]
  Study Week 9: number analyzed (Participants) | 3 | 2
  Study Week 9 | -1.42 [-2.1 to -0.45] | -2.865 [-3.37 to -2.36]
  Study Week 10: number analyzed (Participants) | 2 | 2
  Study Week 10 | -1.58 [-2.47 to -0.69] | -2.62 [-3.3 to -1.94]
  Study Week 11: number analyzed (Participants) | 2 | 2
  Study Week 11 | -1.94 [-2.83 to -1.05] | -2.81 [-3.59 to -2.03]
  Study Week 12: number analyzed (Participants) | 2 | 2
  Study Week 12 | -0.935 [-1.7 to -0.17] | -2.775 [-3.19 to -2.36]

11. Secondary Outcome: Adequacy of Growth as Evaluated by Z-scores for Head Circumference
Description: as for outcome 10
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Median (Full Range); unit: z-score
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 12 | 9
z-score
  Birth | -0.99 [-4.12 to 0.82] | -0.94 [-1.65 to 0.95]
  Study Week 1 | -1.18 [-3.8 to 0.25] | -1.3 [-1.83 to 0.5]
  Study Week 2: number analyzed (Participants) | 11 | 8
  Study Week 2 | -1.36 [-3.91 to 0.04] | -0.82 [-2.31 to -0.02]
  Study Week 3: number analyzed (Participants) | 11 | 6
  Study Week 3 | -1.67 [-3.66 to -0.03] | -1 [-1.58 to 0.17]
  Study Week 4: number analyzed (Participants) | 10 | 5
  Study Week 4 | -1.745 [-2.74 to -0.81] | -1.1 [-1.45 to -0.79]
  Study Week 5: number analyzed (Participants) | 8 | 3
  Study Week 5 | -1.225 [-2.81 to 0.15] | -1.38 [-1.41 to -1.32]
  Study Week 6: number analyzed (Participants) | 7 | 3
  Study Week 6 | -1.34 [-2.77 to 0.23] | -1.56 [-1.74 to -1.18]
  Study Week 7: number analyzed (Participants) | 5 | 2
  Study Week 7 | -0.79 [-1.6 to -0.12] | -1.095 [-1.25 to -0.94]
  Study Week 8: number analyzed (Participants) | 4 | 2
  Study Week 8 | -0.845 [-1.17 to -0.08] | -1.455 [-1.61 to -1.3]
  Study Week 9: number analyzed (Participants) | 3 | 2
  Study Week 9 | -1.44 [-1.49 to -0.24] | -1.39 [-1.51 to -1.27]
  Study Week 10: number analyzed (Participants) | 2 | 2
  Study Week 10 | -0.84 [-1.75 to 0.07] | -1.255 [-1.35 to -1.16]
  Study Week 11: number analyzed (Participants) | 2 | 2
  Study Week 11 | -0.935 [-2.05 to 0.18] | -1.19 [-1.19 to -1.19]
  Study Week 12: number analyzed (Participants) | 2 | 2
  Study Week 12 | -0.63 [-1.15 to -0.11] | -1.31 [-1.88 to -0.74]

12. Secondary Outcome: Adverse Events, as Defined by Any Episode of Sepsis and Catheter-related Blood Stream Infections
Description: The number of episodes were compared between the standard and reduced lipid groups of suspected sepsis episodes, NEC, or catheter-related blood stream infections.
Time Frame: 12 weeks
Population: Subjects who experienced an episode of suspected sepsis, catheter-related blood stream infection, or NEC
Measure: Number; unit: episodes
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 1 | 2
episodes
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 2
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 3
  Participant 3: number analyzed (Participants) | 1 | 0
  Participant 3 | 1 |

13. Secondary Outcome: Bayley Scales for Infant and Toddler Development (BSID-III) at One Year
Description: The Bayley Scales of Infant and Toddler Development (BSID-III) is designed to assess developmental functioning of infants and toddlers, ages 1 month to 42 months. The instrument includes five distinct scales, of which three scales and associated subscales are utilized for the purposes of this study: cognitive, language (receptive and expressive communication) and motor (fine motor and gross motor). Raw scores are converted to scaled scores using age-standardized norm. The cognitive scaled scores range from 1-19. 1 is a low score and 19 is a high score. The Language scaled scores are calculated by adding the Receptive Communication scores ranging from 1-19 and the Expressive communication scores ranging from 1-19 to give the Language Scaled score of 2-38. The Motor scaled scores are calculated by adding the Fine Motor scores ranging from 1-19 and the Gross Motor scores ranging from 1-19 to give the Motor scaled ranging from 2-38. Higher scores are better than lower scores.
Time Frame: 1 year
Population: Participants who returned for their one year follow up
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 5 | 3
scores on a scale
  Cognitive Scaled | 9 [7 to 14] | 10 [9 to 13]
  Language Scaled | 18 [15 to 20] | 16 [13 to 17]
  Motor Scaled | 15 [15 to 20] | 20 [12 to 20]

14. Secondary Outcome: Bayley Scales for Infant and Toddler Development (BSID-III) at Two Years
Description: as for outcome 13
Time Frame: 2 years
Population: Participants who returned for their 2 year follow-up (Note: subjects who did not do their one year follow up were included)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 6 | 2
score on a scale
  Cognitive Scaled | 7.5 [3 to 9] | 10.5 [9 to 12]
  Language Scaled | 17 [4 to 21] | 23 [22 to 24]
  Motor Scaled | 17.5 [9 to 20] | 22 [22 to 22]

15. Secondary Outcome: MacArthur-Bates Communicative Development Inventories (CDI)
Description: The MacArthur-Bates Communicative Development Inventories (CDI) are parent report instruments which capture information about children's developing abilities in early language. Scores are reported as percentiles compared to age-standardized norms. Higher scores are better than lower scores.
Time Frame: 2 years
Population: as for outcome 14
Measure: Median (Full Range); unit: percentile
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 6 | 2
percentile
  Vocabulary Percentile | 25 [7 to 52.5] | 57.5 [42.5 to 72.5]
  Word Forms Percentile | 20 [10 to 65] | 50 [35 to 65]
  Complexity Percentile | 16.25 [7.5 to 77.5] | 88.75 [85 to 92.5]

16. Secondary Outcome: Brief Infant Toddler Social Emotional Assessment (BITSEA) Part 1 of 2
Description: Dichotomous scores are generated based on cut-off scores, which identify subjects to be at risk. The problem scale measures behaviors of the child that if present, represent a problem. The competence scale measures behaviors of the child that if absent, represent a problem. BITSEA percentile rankings are determined from a table that has a limited range and are adjusted for age and sex. A high problem score leads to a low problem percentile. A high competence score leads to a high competence percentile. Percentile rankings for both problem and competence scores range from "4% or less" to "26% or higher". 4 is the lowest percentile score and 26 is the highest percentile score. The 25th percentile is the lower limit of the average range. Higher percentile scores are better than lower percentile scores in both problem and competence categories.
Time Frame: 2 years
Population: as for outcome 14
Measure: Median (Full Range); unit: percentile
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 6 | 2
percentile
  Problem Percentile | 26 [12 to 26] | 26 [26 to 26]
  Competence Percentile | 25.5 [4 to 26] | 26 [26 to 26]

17. Secondary Outcome: Gross Motor Function Classification System (GMFCS)
Description: This classification is based on observation with a scale of 1-5. A lower number classification is better than a higher classification, with 1 being the best.
Time Frame: 2 years
Population: Subjects who were evaluated using the GMFCS.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 5 | 2
Participants
  Subjects with a classification of 1 | 5 | 2
  Subjects with a classification of 2 | 0 | 0
  Subjects with a classification of 3 | 0 | 0
  Subjects with a classification of 4 | 0 | 0
  Subjects with a classification of 5 | 0 | 0

18. Secondary Outcome: Behavioral Assessment System for Children-Third Edition (BASC3) Part 1 of 2
Description: The Behavioral Assessment System for Children-Third Edition is a comprehensive set of forms that helps to understand the behaviors and emotions of children. Scores are reported as T-Scores. T-Scores range from 0-120. In a normative population, the mean of standard scores is 50, and standard deviation is 10. For Externalizing Problems T-Score, Internalizing Problems T-Score, Behavioral Symptoms Index T-Score, Clinical Probability Index T-Score, and Functional Impairment Index T-Score lower scores are better than higher scores. For these categories, higher scores are more problematic with scores between 60-70 regarded as "at risk" and scores 70 and above regarded as clinically significant and requiring further assessment and possible treatment. For Adaptive Skills T-Score, a higher score is better than a lower score. For Adaptive Skills T-Score, lower scores are more problematic with scores between 30-40 regarded as "at risk" and scores at or below 30 regarded as clinically significant.
Time Frame: 2 years
Population: as for outcome 14
Measure: Median (Full Range); unit: T-Score
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 6 | 2
T-Score
  Externalizing Problems T-Score | 43 [38 to 66] | 55.5 [44 to 67]
  Internalizing Problems T-Score | 47 [41 to 56] | 48 [43 to 53]
  Behavioral Symptoms Index T-Score | 48.5 [41 to 65] | 53 [45 to 61]
  Clinical Probability Index T-Score | 51.5 [40 to 69] | 50.5 [40 to 61]
  Functional Impairment Index T-Score | 52 [42 to 61] | 52 [42 to 62]
  Adaptive Skills T-Score | 41 [35 to 51] | 49.5 [42 to 57]

19. Secondary Outcome: Behavioral Assessment System for Children-Third Edition (BASC3) Part 2 of 2
Description: The Behavioral Assessment System for Children-Third Edition is a comprehensive set of forms that helps to understand the behaviors and emotions of children. For Overall Executive Functioning Index, Attentional Control Index, Behavioral Control Index, and Emotional Control Index, scores are "Not Elevated" or "Elevated". Not Elevated is better than Elevated.
Time Frame: 2 years
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 6 | 2
Participants
  Overall Executive Functioning Index: Not Elevated | 5 | 1
  Overall Executive Functioning Index: Elevated | 1 | 1
  Attentional Control Index: Not Elevated | 6 | 1
  Attentional Control Index: Elevated | 0 | 1
  Behavioral Control Index: Not Elevated | 5 | 1
  Behavioral Control Index: Elevated | 1 | 1
  Emotional Control Index: Not Elevated | 5 | 1
  Emotional Control Index: Elevated | 1 | 1

20. Secondary Outcome: Brief Infant Toddler Social Emotional Assessment (BITSEA) Part 2 of 2
Description: Dichotomous scores are generated based on cut-off scores, which identify subjects to be at risk. The problem scale measures behaviors of the child that if present, represent a problem. The competence scale measures behaviors of the child that if absent, represent a problem.
Time Frame: 2 years
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lipid | Standard Lipid
Number analyzed (Participants) | 6 | 2
Participants
  No Problem | 5 | 2
  Possible Problem | 1 | 0
  No Deficit/Delay | 5 | 2
  Possible Deficit/Delay | 1 | 0

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Reduced Lipid | Standard Lipid
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/12 | 4/9
Other Adverse Events (participants affected / at risk) | 8/12 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced Lipid (N=12) | Standard Lipid (N=9)
Sepsis (General disorders) | 0 | 2
PNAC (Hepatobiliary disorders) | 2 | 3
Necrotizing enterocolitis (Infections and infestations) | 1 | 1
PICC associated DVT (Vascular disorders) | 0 | 2
Bowel obstruction (Gastrointestinal disorders) | 1 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ischemic Bowel Disease (Gastrointestinal disorders) | 0 | 1
Hyponatremia (General disorders) | 0 | 1
Acute respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Anemia- Serious (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal Failure- Short Bowel Syndrome (Gastrointestinal disorders) | 0 | 1
Inadequate Weight Gain (General disorders) | 0 | 1
Metabolic Acidosis- normal anion gap and bicarbonate loss (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced Lipid (N=12) | Standard Lipid (N=9)
Line Complication, Removal, or Replacement (Surgical and medical procedures) | 4 | 2
Bradycardia with Tachypnea (General disorders) | 0 | 1
Hyperglycemia (General disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Hypertension (General disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oral Thrush (Infections and infestations) | 1 | 0
Non-severe Anemia (General disorders) | 0 | 1
Inadequate weight gain- non-severe (General disorders) | 1 | 0
Enteritis (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
There was a smaller sample size than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT02357576/Prot_SAP_000.pdf